CLINICAL TRIAL: NCT06506773
Title: A Natural History Study of Exocrine Pancreatic Function in Infants With Cystic Fibrosis Less Than 12 Months of Age
Brief Title: Natural History Study of Exocrine Pancreatic Function in Infants With Cystic Fibrosis (CF)
Status: Completed | Type: Observational
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: VX24-445-130
Record Dates: First submitted 2024-06-27; First posted 2024-07-17 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort A: Observational follow-up study to characterize the natural history of exocrine pancreatic function by measuring FE-1 in infants with CF.

SUMMARY:
The purpose of the study is to evaluate the natural history of exocrine pancreatic function by assessing Fecal elastase-1 (FE-1) in infants with CF during their first year of life.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with CF less than (<) 6 months of age at the index date
* Participants not eligible to receive commercial Kalydeco™ (based on local product labels) and are not receiving Kalydeco or any other cystic fibrosis transmembrane conductance regulator gene (CFTR) modulator

Key Exclusion Criteria:

* Participant whose mother took any CFTR modulator while pregnant with the participant, or who has any history of exposure to a CFTR modulator

Other protocol defined Inclusion/Exclusion criteria apply.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with CF less than (<) 6 months of age at the index date who are not eligible for commercial Kalydeco™ (according to local product labels). The day of enrollment into this study will be referred to as the "index date".
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants with FE-1 greater than or equal to (≥) 200 microgram per gram (µg/g) Over Time | From Enrollment up to the Infant turning 12 Months of Age

SECONDARY OUTCOMES:
FE-1 level Over Time | From Enrollment up to the Infant turning 12 Months of Age

CONTACTS AND LOCATIONS:
Locations (50):
- United States (22):
  - Johns Hopkins All Children's Hospital Outpatient Care Center, St. Petersburg, Florida
  - St. Luke's Cystic Fibrosis Center of Idaho, Boise, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Boston Childrens Hospital, Boston, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - Children's Respiratory and Critical Care Specialists, P.A., Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Billings Clinic, Billings, Montana
  - Children's Nebraska, Omaha, Nebraska
  - Duke University Medical Center, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Toledo Children's Hospital/Pediatric Pulmonary & Cystic Fibrosis Center, Toledo, Ohio
  - Prisma Health Clinical Research Unit - Midlands, Columbia, South Carolina
  - Sanford Children's Speciality Clinic, Sioux Falls, South Dakota
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - Virginia Commonwealth University Hospital Systems, Children's Pavilion, Richmond, Virginia
  - Providence Pediatric Pulmonary & Cystic Fibrosis Clinic, Spokane, Washington
  - West Virginia University, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - The Kids Research Institute Australia, Nedlands
  - Women's and Children's Hospital, North Adelaide
  - Queensland Children's Hospital, South Brisbane
- Canada (4):
  - McGill University Health Centre, Glen Site, Montreal Children's Hospital, Montreal
  - Centre Hospitalier de Quebec - Universite Laval, Québec
  - The Hospital for Sick Children, Toronto
  - British Columbia Children's Hospital, Vancouver
- Fakultni nemocnice v Motole, Prague, Czechia
- Germany (3):
  - Charite Paediatric Pulmonology Department, Berlin
  - Kinderklinik III, Abt. fur Pneumologie, Essen
  - Klinikum Westbrandenburg (CF), Potsdam
- Azienda Ospedaliero Universitaria Ospedale Pediatrico Meyer, Florence, Italy
- New Zealand (2):
  - Canterbury District Health Board, Christchurch
  - Starship Children's Hospital, Grafton
- Pediatric Hospital Polanki named of Maciej Płażyński, Gdansk, Poland
- Spain (3):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Kinderspital Zurich, Zurich, Switzerland
- United Kingdom (9):
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol Royal Hospital for Children, Bristol
  - Royal Hospital for Children, Glasgow
  - Leeds Regional Children's Cystic Fibrosis Centre, Leeds
  - Leicester Royal Infirmary, University of Leicester, Leicester
  - Great Ormond Street Hospital for Children, London
  - The Royal London Children's Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Nottingham University Hospitals NHS Trust, Children's Clinical Research Facility, Nottingham
  - Royal Stoke University Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https: https://www.vrtx.com/our-science/clinical-trials-data-sharing/